CLINICAL TRIAL: NCT07065240
Title: A Randomized, Parallel-Group, Double-Blind, Placebo-Controlled, Monotherapy Study of the Efficacy, Safety, and Tolerability of SPT-300 in Adults With Major Depressive Disorder (MDD), With or Without Anxious Distress
Brief Title: A Study to Evaluate the Efficacy and Safety of SPT-300 (GlyphAllo) in Participants With Major Depressive Disorder, With or Without Anxious Distress (BUOY-1 Study)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seaport Therapeutics (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPT-300-2024-203; 2025-521240-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD); Major Depressive Disorder With Anxious Distress
Keywords: Major Depressive Disorder; Depressive Disorder; Depression; Anxiety; Mood Disorders; BUOY-1 Study; SPT-300; LYT-300; GlyphAllo; Glyph Allopregnanolone
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder; Depression; Anxiety Disorders; Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SPT-300 (Experimental): Participants will receive SPT-300 capsules once daily for 42 days
  Interventions: Drug: SPT-300
- Placebo (Placebo Comparator): Participants will receive matching placebo once daily for 42 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPT-300 — A prodrug of allopregnanolone, a small molecule drug
  Other Names: LYT-300; GlyphAllo; Glyph Allopregnanolone
  Arms: SPT-300
Drug: Placebo — Placebo for SPT-300
  Arms: Placebo

SUMMARY:
This is a randomized, parallel-group, double-blind, placebo-controlled, monotherapy study to evaluate the efficacy, safety, and tolerability of SPT-300 (GlyphAllo) in adults with major depressive disorder (MDD), with or without anxious distress.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female between 18 and 65 years of age, inclusive willing and able and have capacity to provide written informed consent.
* Participants must have a primary diagnosis of MDD. Participants with a diagnosis of comorbid generalized anxiety disorder, social anxiety disorder, or panic disorder (with or without agoraphobia) may be included if not the focus of treatment over the past 6 months prior to Screening and the Investigator considers MDD to be the primary diagnosis at Screening and Baseline.
* Eligible participants must have a current depressive episode of at least 4 weeks, but no greater than 18 months in duration prior to Screening.
* Women of childbearing potential (WOCP) must not plan to become pregnant during the course of the study or be currently breastfeeding. WOCP agree to use an acceptable form of highly effective contraception during participation in the study and for 30 days after receiving the last dose of study treatment.
* Body mass index (BMI) between 18 to 40 kg/m2, inclusive.
* Participant is willing and able to refrain from the use of drugs of abuse.

Exclusion Criteria:

* History of, or current presentation consistent with:

  1. any depressive episode with psychotic or catatonic features.
  2. any bipolar manic, hypomanic or mixed episode, and substance-induced (e.g., antidepressant-induced) manic, hypomanic/mixed episode.
  3. bipolar disorder, including history of bipolar depression, or current presentation consistent with bipolar depression.
  4. schizophrenia, schizoaffective, or other psychotic disorder.
  5. obsessive-compulsive disorder.
  6. any persistent neurocognitive disorder.
* History of treatment-resistant depression defined as 2 or more failed treatments of adequate dose and duration in the current depressive episode.
* Psychiatric hospitalization within current depressive episode.
* Evidence or history of clinically significant diseases which can affect the patients' participation.
* Previous history of intolerance or significant adverse effects, including drug allergy to allopregnanolone or any components of the SPT-300/placebo formulation.
* Participant has a history of drug or alcohol use disorder.
* Participants with a positive test for cannabinoids.
* Clinically significant risk of suicide or harm to self or others.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline to Day 42 in Hamilton Depression Rating Scale-17 (HAM-D-17) Total Score | Baseline (Day 0) to Day 42
  HAM-D-17 is a 17-item, clinician-administered rating scale to assess the severity of symptoms in participants diagnosed with depression. The HAM-D-17 comprises individual ratings related to the following symptoms: depressed mood (sadness, hopeless, helpless, worthless), feelings of guilt, suicide, insomnia (early, middle, late), work and activities, retardation (slowness of thought and speech; impaired ability to concentrate; decreased motor activity), agitation, anxiety (psychic and somatic), somatic symptoms (gastrointestinal and general), genital symptoms, hypochondriasis, loss of weight, and insight. HAM-D Total Scores range from 0 to 52, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Change From Baseline to Day 42 in Clinical Global Impression - Severity (CGI-S) | Baseline (Day 0) to Day 42
  The CGI-S is a clinician-administered rating scale to assess the severity of the participant's illness at the time of the assessment relative to the clinician's past experience with patients who have the same diagnosis. Scores range from 1 to 7, with higher scores indicating more severe illness.

CONTACTS AND LOCATIONS:
Overall Officials: David Walling, Ph.D., Principal Investigator — Collaborative Neuroscience Research - Garden Grove
Locations (39):
- United States (16):
  - Seaport Investigator Site, Chino, California
  - Seaport Investigator Site, Garden Grove, California
  - Seaport Investigator Site, Glendale, California
  - Seaport Investigator Site, Cromwell, Connecticut
  - Seaport Investigator Site, West Palm Beach, Florida
  - Seaport Investigator Site, Atlanta, Georgia
  - Seaport Investigator Site, Decatur, Georgia
  - Seaport Investigator Site, Marietta, Georgia
  - Seaport Investigator Site, Boston, Massachusetts
  - Seaport Investigator Site, St Louis, Missouri
  - Seaport Investigator Site, Brooklyn, New York
  - Seaport Investigator Site, New York, New York
  - Seaport Investigator Site, Staten Island, New York
  - Seaport Investigator Site, Independence, Ohio
  - Seaport Investigator Site, North Canton, Ohio
  - Seaport Investigator Site, Irving, Texas
- Bulgaria (2):
  - Seaport Investigator Site, Plovdiv
  - Seaport Investigator Site, Sofia
- Czechia (3):
  - Seaport Investigator Site, Brno
  - Seaport Investigator Site, Pilsen
  - Seaport Investigator Site, Prague
- Germany (4):
  - Seaport Investigator Site, Berlin, Brandenburg
  - Seaport Investigator Site, Schwerin, Mecklenburg-Vorpommern
  - Seaport Investigator Site, Bad Homburg
  - Seaport Investigator Site, Chemnitz
- Poland (11):
  - Seaport Investigator Site, Bełchatów
  - Seaport Investigator Site, Bialystok
  - Seaport Investigator Site, Bydgoszcz
  - Seaport Investigator Site, Gdansk
  - Seaport Investigator Site, Katowice
  - Seaport Investigator Site, Leszno
  - Seaport Investigator Site, Poznan
  - Seaport Investigator Site, Torun
  - Seaport Investigator Site, Tuszyn
  - Seaport Investigator Site, Warsaw
  - Seaport Investigator Site, Wroclaw
- Slovakia (3):
  - Seaport Investigator Site, Bratislava
  - Seaport Investigator Site, Rimavská Sobota
  - Seaport Investigator Site, Vranov nad Topľou